CLINICAL TRIAL: NCT05864573
Title: A Phase 1 Dose Escalation, Tolerability, Safety and Pharmacokinetics Study of ZGGS15 in Patients With Advanced Solid Tumors
Brief Title: Study of ZGGS15 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGGS15-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZGGS15 (Experimental)
  Interventions: Biological: ZGGS15

INTERVENTIONS:
Biological: ZGGS15 — ZGGS15 for dose escalations are set as 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, and 30 mg/kg, intravenous infusion, once every 3 weeks.

SUMMARY:
This is a multi-center, open-label, Phase 1 clinical study of ZGGS15 for the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female, 18-70 years of age;
* Histologically or cytologically confirmed diagnosis of advanced solid tumors, in whom the available standard treatments failed;
* Must have at least 1 measurable lesion per RECIST v1.1;
* Eastern Cooperative Oncology Group performance status of 0 or 1;
* Life expectancy ≥ 3 months;
* All adverse events from prior treatment have either returned to baseline or CTCAE v5.0≤Grade 1;
* Both male and female participants (unless postmenopausal, surgical sterilization) and partners must agree to use a reliable form of contraception during the study treatment period and for at least 6 months after the last dose of the study drug.

Exclusion Criteria:

* Medical history, computed tomography (CT) or magnetic resonance imaging (MRI) results indicate the existence of the central nervous system (CNS) metastases；
* Uncontrollable third cavity effusion requiring repeated drainage, which was judged by the investigator to be unsuitable for study;
* The main organ function meets any of the following criteria within 7 days prior to treatment:

  * Hematological function: absolute neutrophil count (ANC) < 1.5 × 10^9/L, platelet (PLT) < 75 × 10^9/L, or hemoglobin (Hb) < 100 g/L;
  * Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 × upper limit of normal (ULN), ALT and AST ≥ 5×ULN for patients with liver metastases; total bilirubin (TBIL) ≥ 1.5×ULN; albumin < 30 g/L;
  * Blood cholesterol > 300 mg/dL or > 7.75 mmol/L;
  * Creatinine clearance (Cockcroft-Gault formula) < 50 mL/min;
  * International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (APTT) > 1.5×ULN;
* Any other malignancy within 5 years;
* Abnormal thyroid function with clinical symptoms or diabetes, which cannot be controlled by available treatments;
* History of autoimmune disease, including but not limited to systemic lupus erythematosus, nephritis, psoriasis, rheumatoid arthritis, inflammatory bowel disease, autoimmune hepatitis;
* Previous immune checkpoint inhibitors induced ≥ Grade 2 immune-related adverse reactions in vital organs, including but not limited to myocarditis and central nervous system toxicity; rapidly tumor progressed after previous PD-1 inhibitor treatment;
* Interstitial lung disease, non-infectious pneumonitis, and radiation-induced pneumonia with symptoms and/or requiring steroids for treatment;
* Received prior allogeneic stem cell transplantation or solid organ transplantation;
* Active infection within 1 week before the first administration currently requires systemic anti-infective therapy;
* Known allergy to other mAbs or any antibody excipient, severe allergic reaction to humanized antibodies or fusion proteins, and history of anaphylactoid reaction or other hypersensitivity reactions;
* Known history of diagnosed neurological or mental disorders, for example, epilepsy, dementia, etc.;
* Patients were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLTs) | Up to 21Days
  A DLT is defined as any of the following adverse events occurring from the first dose to the end of the first Cycle (21 days), unless the investigator deems that the AE is clearly related to the disease progression or definitely due to an external cause.
The maximum tolerated dose (MTD) | Up to 24 Months
  During the dose-escalation stage, if ≥ 2 patients in a dose group experienced DLTs, then the dose level will be considered to be an intolerable dose, and the previous lower dose will be considered to be the MTD.
The recommended dose for subsequent study | Up to 24 Months
  The recommended dose for the subsequent study will be based on the data of preliminary efficacy, safety, PK, receptor occupancy results and biomarker (for example, immune activation), etc. from the dose-escalation phase, and will be fully evaluated among the investigators and the sponsor. The recommended dose for subsequent study should have at least 6 evaluable patients.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 Months
  Disease control rate (DCR) will be determined from investigator derived tumor assessments per RECIST v. 1.1.
Duration of response (DOR) | Up to 24 Months
  Objective Response Rate will be determined from investigator derived tumor assessments per RECIST v. 1.1.
Disease control rate (DCR) | Up to 24 Months
  Disease control rate (DCR) will be determined from investigator derived tumor assessments per RECIST v. 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China